CLINICAL TRIAL: NCT02830919
Title: Phase III Clinical Study, Multicenter, Randomized, Single-blind, Parallel Groups for Safety Evaluation and Non-inferiority of Efficacy of Glucosamine Sulfate Plus Chondroitin Sulfate From Bovine Origin (Eurofarma Laboratorios S.A.) Versus Condroflex ® in the Treatment of Symptomatic Knee Primary Osteoarthritis
Brief Title: Clinical Study of Non-inferiority With Participants Diagnosed With Primary Knee OA (GLACIAL)
Acronym: GLACIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF140
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis of knee; Glucosamine sulfate; Chondroitin sulfate
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucosamine and chondroitin sulfate combination (Eurofarma) (Experimental): Glucosamine sulfate 1500mg plus chondroitin sulfate 1200mg combination, manufactured by Eurofarma Laboratórios S.A., administered once a day for 24 weeks.
  Interventions: Drug: Glucosamine and chondroitin sulfate combination (Eurofarma)
- Glucosamine and chondroitin sulfate combination (Zodiac) (Active Comparator): Glucosamine sulfate 1500mg plus chondroitin sulfate 1200mg combination, manufactured by Zodiac Produtos Farmacêuticos S.A. (Condroflex®), administered once a day for 24 weeks.
  Interventions: Drug: Glucosamine and chondroitin sulfate combination (Zodic)

INTERVENTIONS:
Drug: Glucosamine and chondroitin sulfate combination (Eurofarma)
  Arms: Glucosamine and chondroitin sulfate combination (Eurofarma)
Drug: Glucosamine and chondroitin sulfate combination (Zodic)
  Arms: Glucosamine and chondroitin sulfate combination (Zodiac)

SUMMARY:
This phase III clinical study will be conducted in Brazilian research sites. It will be included in the study 314 participants diagnosed with primary knee OA according to the classification criteria of the ACR. After a washout period, the participants will be randomized to receive the combination of glucosamine sulfate + chondroitin sulfate of bovine origin of Eurofarma Laboratorios S.A. (N= 157) or the combination of glucosamine sulfate + chondroitin sulfate of Zodiac Pharmaceuticals S.A. Condroflex ® (N = 157). The treatment period of the study will be of 24 weeks. Each participant will perform seven visits to the research site. The main evaluations will be the improve of pain in the target knee by questionnaire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and quality of life by SF-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients meeting all the following criteria will be enrolled in the study:

1. Aged ≥ 40 years.
2. Clinical and radiological diagnosis of primary (idiopathic) arthrosis of knee according to the criteria of the American College of Rheumatology (ACR).
3. Kellgren and Lawrence radiological classification of degree 2 or 3 in x-ray of knee-target obtained in 3 months prior to the screening visit of the study.
4. Presence of painful symptoms in the target knee in the last 3 months due to osteoarthritis.
5. Visual analogue scale for evaluation of the pain of osteoarthritis of knee by the research participant in the screening visit ≥ 40 mm
6. Average score ≥ 40 mm in the subscale of "pain" (from 0 to 100 mm) in the target knee of the questionnaire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), in the randomization visit.
7. Functional class ACR from I to III.
8. Signing the Informed Consent Form (ICF) before the performance of any study procedure.

Exclusion Criteria:

Patients meeting at least one of the following criteria will be excluded from the study:

1. Diagnosis of septic arthritis, inflammatory arthritis (as rheumatoid arthritis), gout, pseudogout, Paget's disease, dysplasias or congenital joint abnormalities.
2. Presence of inflammatory signals (edema, erythema or joint effusion) in the target knee, considered to be clinically significant by investigator.
3. Serious target knee joint misalignment, defined by investigator.
4. Predominantly patellofemoral Osteoarthritis in the target knee.
5. Historical of severe trauma or surgery (including arthroscopy) in the target knee in the 6 months before the screening visit.
6. Planned Surgery to the target knee
7. Symptomatic Osteoarthritis of the ipsilateral hip.
8. Use of non-steroidal anti-inflammatory, dipyrone and opioid analgesics or narcotics from the screening visit, or a washout period for these medicines less than those defined by the Protocol, before the randomization visit .
9. Oral Glucocorticoids, intravenously or intramuscularly in the 30 days prior to the screening visit.
10. Intraarticular corticosteroid Injection and/or hyaluronic acid in the target knee in 6 months prior to the screening visit.
11. Use of the following drugs in the periods described below, before the screening visit:

    1. Diacerein, chloroquine or soybean and avocado unsaponifiables extracts in the last 3 months.
    2. Duloxetine hydrochloride in the last 30 days.
    3. Glucosamine Sulphate and/or chondroitin sulfate in the last 6 months.
    4. Strontium ranelate for the past 6 months.
12. Historical of allergy or intolerance to treatment of the study or to paracetamol.
13. Physiotherapy or irregular practice of physical activity beginning in the 3 months prior to the screening visit.
14. Diagnosis of fibromyalgia, collagenosis or significative vascular/neurologica diseases in lower limbs that may confuse the analysis of the study.
15. Body mass index ≥ 40 kg/m2.
16. Need to use cane, crutches or a walker.
17. Presence of infectious hepatitis active or history of hepatitis medicinal products.
18. Results of ALT, AST and total bilirubin and fractions above the upper limit of normal.
19. Serum creatinine level above the upper limit of normal.
20. Fasting blood glucose > 110 mg/dL or glycated hemoglobin > 6.5%.
21. Use of anticoagulants.
22. Consumption of alcohol more than one dose a day (women) or two doses a day (men).
23. Presence of serious diseases or not controlled.
24. Planned surgery to occur during the period of participation in the study.
25. Presence of pregnancy or breastfeeding.
26. Women of childbearing potential must agree to use highly effective contraception.
27. Participation in a clinical trial protocol within the previous 12 months unless, at the investigator's discretion, his or her participation may imply a direct benefit for the participant.
28. Presence of any condition which, at the investigator's discretion, may consider the participation of the patient inadequate for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Absolute change of pain WOMAC subscale score 24 weeks after initiation of treatment. | 24 weeks

SECONDARY OUTCOMES:
Absolute change the overall assessment of the disease by the investigator along treatment as measured by Visual Analog Scale from 0 to 100mm. | 24 weeks
Absolute change score of physical and mental components of the questionnaire SF-12 24 weeks after initiation of treatment compared to baseline. | 24 weeks
Incidence and profile of adverse events coded as MedDRA by treatment group. | 24 weeks
Frequency of treatment discontinuation for adverse events and laboratory abnormalities. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Goiânia, Goiás
  - Curitiba, Paraná
  - Maringá, Paraná
  - São Paulo, São Paulo

REFERENCES:
- [Derived] Lomonte ABV, Gimenez E, da Silva AC, Radominski SC, Scheinberg MA, Ximenes AC, de Freitas Zerbini CA. Treatment of knee osteoarthritis with a new formulation of a fixed-dose combination of glucosamine sulfate and bovine chondroitin: a multicenter, randomized, single-blind, non-inferiority clinical trial. Adv Rheumatol. 2021 Jan 19;61(1):7. doi: 10.1186/s42358-021-00165-9. PMID 33468249